CLINICAL TRIAL: NCT02093741
Title: ADVATE 2 mL (Reconstituted in 2 mL SWFI) POST-AUTHORIZATION SAFETY SURVEILLANCE STUDY
Brief Title: ADVATE 2 mL Post-Authorization Safety Surveillance (PASS)
Status: Completed | Type: Observational
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: 061101
Record Dates: First submitted 2014-03-19; First posted 2014-03-21 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Hemophilia A; Congenital Factor VIII (FVIII) Deficiency
MeSH Terms: conditions — Hemophilia A | interventions — F8 protein, human; Factor VIII

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ADVATE - 2mL
  Interventions: Biological: Octocog alfa (recombinant human coagulation factor VIII) [ADVATE]

INTERVENTIONS:
Biological: Octocog alfa (recombinant human coagulation factor VIII) [ADVATE] — The investigators shall determine all treatment regimens according to product labeling information and standard practice.
  Other Names: Antihemophilic Factor (Recombinant)- Plasma/albumin free method (rAHF-PFM); ADVATE

SUMMARY:
This is a Post-Authorization Safety Surveillance (PASS) study designed to collect data on the safety and effectiveness of ADVATE reconstituted in 2 mL Sterile water for injection (SWFI) during routine clinical practice in children until 12 years of age. This surveillance study is a post-licensure commitment for ADVATE reconstituted in 2 mL SWFI.

ELIGIBILITY:
Inclusion Criteria:

* Severe or moderately severe hemophilia A (baseline Factor VIII (FVIII) ≤ 2%)
* ≤12 years of age
* Participant's legally authorized representative(s) has provided written informed consent
* Participant is prescribed ADVATE and will only receive ADVATE reconstituted in 2 mL sterile water for injection (SWFI)
* Documented history of prior exposure to ADVATE
* Documented evidence of negative inhibitor test result during ≤10 EDs prior to study entry

Exclusion Criteria:

* Known hypersensitivity to the active substance or to any of the excipients
* Known allergic reaction to mouse or hamster proteins
* Participant has a requirement for a major surgical procedure at the time of enrollment
* Participant has no prior exposure to a FVIII concentrate
* Participant currently being treated with an immune tolerance induction (ITI) regimen
* Participant has been diagnosed with an inherited or acquired hemostatic defect other than hemophilia A (eg, qualitative platelet defect or von Willebrand disease)
* Participant has participated in another clinical study involving an investigational product (IP) or investigational device within 30 days prior to enrollment or is scheduled to participate in another clinical study involving an IP or investigational device or PASS registry during the course of this study

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will include 60 evaluable participants aged = 12 years with severe or moderately severe hemophilia A (Factor VIII (FVIII) = 2%) with documented prior exposure to FVIII concentrates.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2013-09-20 (Actual); Primary Completion 2016-01-20 (Actual); Study Completion 2016-01-20 (Actual)

PRIMARY OUTCOMES:
Incidence of all local and general, hypersensitivity and infusion-related reactions, irrespective of product-related causality for the adverse events (AEs). | 6 months

SECONDARY OUTCOMES:
Number and type of adverse events (or adverse experiences) (AEs) considered by the investigator to be causally related to ADVATE reconstituted in 2 mL sterile water for injection (SWFI) | 6 months
  Causally related = possibly or probably related
Number of Factor VIII (FVIII) inhibitors in all participants | 6 months
Number of Factor VIII (FVIII) inhibitors in Previously Treated Patients (PTPs) (> 50 Exposure Days (EDs)) with baseline Factor VIII (FVIII) < 1% and no history of FVIII inhibitors prior to study entry | 6 months
Number of Factor VIII (FVIII) inhibitors in Previously Treated Patients (PTPs) (> 50 Exposure Days (EDs)) with baseline Factor VIII (FVIII) ≤ 2% and no history of FVIII inhibitors prior to study entry | 6 months
Subjective hemostatic effectiveness rating of excellent, good, fair, or none for each bleeding episode treated | 6 months
Number of bleeding episodes treated with 1, 2, 3, ≥ 4 infusions of ADVATE reconstituted in 2 mL sterile water for injection (SWFI) | 6 months
Total units of ADVATE reconstituted in 2 mL sterile water for injection (SWFI) administered to treat each bleeding episode | 6 months
Overall effectiveness of prophylaxis in participants who are on a prophylactic regimen | 6 months
Global assessment rating of hemostatic effectiveness of ADVATE reconstituted in 2 mL sterile water for injection (SWFI) in surgical or dental procedures | 6 months
  Global assessment rating = excellent, good, fair, or none
Change in Factor VIII (FVIII) treatment satisfaction and preference ratings from caregiver between ADVATE reconstituted in 5 mL and 2 mL sterile water for injection (SWFI) | 6 months
Change in Factor VIII (FVIII) infusion volume and time to mix and infuse FVIII treatment between ADVATE reconstituted in 5 mL and 2 mL sterile water for injection (SWFI) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (17):
- France (8):
  - CHRU Pellegrin, Hématologie - CRTH, Bordeaux
  - Centre Hospitalier Générale, CTH, Chambéry
  - CRTH Laboratoire d'Hématologie CHRU - Hôpital du Bocage, Dijon
  - American Memorial Hospital, Service de Pédiatrie, Reims
  - CHU de Rennes Hôpital Pontchaillou, Rennes
  - Hôpital Nord, Pédiatrie, Saint-Priest-en-Jarez
  - CHRU Purpan, CRTH - Pavillon Sénac, Toulouse
  - CHU de Nancy - Hôpital de Brabois- CRTH - Laboratoire Hémato-Hémostase, Vandœuvre-lès-Nancy
- Germany (2):
  - Universitätskliniken des Saarlandes, Klinik für pädiatrische Onkologie und Hämatologie, Homburg, Saarland
  - Klinikum Stuttgart, Olgahospital, Pädiatrie 5, Stuttgart
- Hungary (4):
  - Heim Pál Children's Hospital, Department of Oncology, Budapest
  - Borsod-Abaúj-Zemplén County Hospital, Pediatric Dep, Miskolc
  - Mohacsi Korhaz, Department of Pediatrics, Mohács
  - Josa Andras Egyetemi Oktatokorhaz, Department of Pediatrics, Nyíregyháza
- United Kingdom (3):
  - Leeds General Infirmary, Leeds, West Yorkshire
  - Birmingham Children's Hospital NHS Trust, Birmingham
  - Great Ormond Street Hospital for Children NHS Trust, London

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/5f6b5fc24db2bf003ab457db